CLINICAL TRIAL: NCT02202811
Title: Circadian Rhythms and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Saurabh Thosar, Saurabh S. Thosar, PhD, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OSA 00010101
Record Dates: First submitted 2014-07-17; First posted 2014-07-29 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Obstructive Sleep Apnea (Experimental): Forced Desynchrony, OSA
  Interventions: Behavioral: Forced Desynchrony
- Control (Placebo Comparator): Forced Desynchrony, Control
  Interventions: Behavioral: Forced Desynchrony

INTERVENTIONS:
Behavioral: Forced Desynchrony — all sleep opportunities and other activities will be scheduled by the experimenter so that by the end of the study these activities are spread evenly across all phases of the internal body clock.

SUMMARY:
The purpose of this study is to understand how behaviors and the effects of the body's internal clock (called the circadian pacemaker) affect the control of the heart and blood pressure.

People with Obstructive Sleep Apnea (OSA) are hypothesized to have altered circadian amplitudes in certain key indices of cardiovascular (CV) and an abnormally advanced circadian phase in some of the same key indices of CV risk. The investigators hypothesize that such changes, taken together, may explain the different timing of heart attack and sudden cardiac death in OSA.

ELIGIBILITY:
* BMI less than 40
* Moderate to severe OSA (AHI)>15
* No current or previous pharmacological treatment for hypertension

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Primary dependent variable: Circadian rhythm amplitude of plasma epinephrine concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma epinephrine concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma epinephrine concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma epinephrine concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Primary dependent variable: Circadian rhythm amplitude of plasma epinephrine reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma epinephrine concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma epinephrine reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma epinephrine concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of plasma epinephrine reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma epinephrine concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma epinephrine reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma epinephrine concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of blood pressure (BP) | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of systolic and diastolic BP during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of blood pressure (BP) | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of systolic and diastolic BP during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Primary dependent variable: Circadian rhythm amplitude of blood pressure (BP) reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in systolic and diastolic BP from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of blood pressure (BP) reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in systolic and diastolic BP from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of blood pressure (BP) reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in systolic and diastolic BP from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of blood pressure (BP) reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in systolic and diastolic BP from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of plasma cortisol concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma cortisol concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma cortisol concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma cortisol concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Primary dependent variable: Circadian rhythm amplitude of plasma cortisol reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma cortisol concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma cortisol reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma cortisol concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of plasma cortisol reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma cortisol concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of plasma cortisol reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma cortisol concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of heart rate | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of heart rate during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of heart rate | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of heart rate during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Primary dependent variable: Circadian rhythm amplitude of heart rate reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in heart rate from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of heart rate reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in heart rate from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of heart rate reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in heart rate from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of heart rate reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in heart rate from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of cardiac vagal tone | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of cardiac vagal tone during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of cardiac vagal tone | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of cardiac vagal tone during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Primary dependent variable: Circadian rhythm amplitude of cardiac vagal tone reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in cardiac vagal tone from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of cardiac vagal tone reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in cardiac vagal tone from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm amplitude of cardiac vagal tone reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in cardiac vagal tone from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Primary dependent variable: Circadian rhythm phase of cardiac vagal tone reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in cardiac vagal tone from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.

SECONDARY OUTCOMES:
Secondary dependent variable: Circadian rhythm amplitude of plasma tissue plasminogen activator inhibitor (tPA) concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma tPA concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma tPA concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma tPA concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Secondary dependent variable: Circadian rhythm amplitude of plasma tPA reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma tPA concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma tPA reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma tPA concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma tPA reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma tPA concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma tPA reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma tPA concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of vascular endothelial function | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of vascular endothelial function during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of vascular endothelial function | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of vascular endothelial function during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Secondary dependent variable: Circadian rhythm amplitude of vascular endothelial function reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in vascular endothelial function from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of vascular endothelial function reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in vascular endothelial function from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of vascular endothelial function reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in vascular endothelial function from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of vascular endothelial function reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in vascular endothelial function from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma plasminogen activator inhibitor 1 (PAI-1) concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma PAI-1 concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma PAI-1 concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma PAI-1 concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Secondary dependent variable: Circadian rhythm amplitude of plasma PAI-1 reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma PAI-1 concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma PAI-1 concentration reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma PAI-1 concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma PAI-1 reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma PAI-1 concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma PAI-1 reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma PAI-1 concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma MDA concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma MDA concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma MDA concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma MDA concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Secondary dependent variable: Circadian rhythm amplitude of plasma MDA reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma MDA concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma malondialdehyde (MDA) reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma MDA concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma MDA concentration reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma MDA concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma malondialdehyde (MDA) reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma MDA concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma 8-isoprostane concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of plasma 8-isoprostane concentration during resting baseline conditions. Circadian rhythm amplitude will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma 8-isoprostane concentration | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian phase of plasma 8-isoprostane concentration during resting baseline conditions. Circadian rhythm phase will be assessed by cosinor analysis of all resting measurements obtained throughout the protocol assessed under constant conditions but at varied circadian phases and stated in relation to the reported habitual sleep time.
Secondary dependent variable: Circadian rhythm amplitude of plasma 8-isoprostane reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma 8-isoprostane concentration from resting baseline to end of 15 minutes of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma 8-isoprostane reactivity to exercise | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma 8-isoprostane concentration from resting baseline to end of 15 minute of steady-state bicycle exercise. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by exercise obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm amplitude of plasma 8-isoprostane reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma 8-isoprostane concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.
Secondary dependent variable: Circadian rhythm phase of plasma 8-isoprostane reactivity to change in posture | Over 5 days
  Comparisons will be made between participants with obstructive sleep apnea (OSA) and healthy controls of the circadian amplitude of change in plasma 8-isoprostane concentration from resting supine to end of 5 minutes of standing. Circadian rhythm amplitude of reactivity will be assessed by cosinor analysis of all changes induced by change in posture obtained throughout the protocol assessed under constant conditions but at varied circadian phases.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Shea, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thosar SS, Bowles NP, Butler MP, McHill AW, Rice SPM, Emens JS, Shea SA. Endogenous Circadian System Attenuates Nighttime Vascular Endothelial Function in People With Untreated Obstructive Sleep Apnea. J Am Heart Assoc. 2025 Nov 18;14(22):e043596. doi: 10.1161/JAHA.125.043596. Epub 2025 Nov 6. PMID 41195783
- [Derived] Thosar SS, Berman AM, Herzig MX, McHill AW, Bowles NP, Swanson CM, Clemons NA, Butler MP, Clemons AA, Emens JS, Shea SA. Circadian Rhythm of Vascular Function in Midlife Adults. Arterioscler Thromb Vasc Biol. 2019 Jun;39(6):1203-1211. doi: 10.1161/ATVBAHA.119.312682. PMID 31070470